CLINICAL TRIAL: NCT05980767
Title: Short Duration Electrical Stimulation to Improve Outcomes After Cubital Tunnel Release (SELECT) Trial
Acronym: SELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Epineuron Technologies Inc. (Industry)
Collaborators: Federal Economic Development Agency for Southern Ontario (FedDev Ontario) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EPNR-CIP-003
Record Dates: First submitted 2023-07-14; First posted 2023-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Neuropathy;Peripheral
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Intervention (Active Comparator): Standard of care plus therapy, which consists of a single, 1 hour dose of electrical stimulation.
  Interventions: Device: Temporary Peripheral Nerve Stimulation System
- Control (No Intervention): Standard of care only.

INTERVENTIONS:
Device: Temporary Peripheral Nerve Stimulation System — Single use medical device. Therapy consists of single, 1 hour dose of electrical stimulation.
  Arms: Experimental Intervention

SUMMARY:
A novel temporary peripheral nerve stimulation system that delivers electrical stimulation therapy in a cubital tunnel release model will be evaluated for feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Ulnar neuropathy at the elbow

Exclusion Criteria:

* Peripheral neuropathy outside of nerve of interest
* Patients with any active implanted device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Eligibility Rate | 1.5 years
  Evaluation of study feasibility through the number of participants who pass all pre-operative screening eligibility criteria
Recruitment Rate | 1.5 years
  Evaluation of study feasibility through the number of participants who complete informed consent and are randomized into a study arm
Retention Rate | 1.5 years
  Evaluation of study feasibility through the number of participants who complete all study activities

OTHER OUTCOMES:
Electromyography (EMG) Denervation Absence/Presence | 1.5 years
  Measurement of electrical activity of a muscle
Nerve Conduction Study (NCS) | 1.5 years
  Measurement of speed of electrical impulse through a nerve
Semmes-Weinstein Monofilament Test | 1.5 years
  Evaluation of sensory recovery through the measurement of a pressure detection threshold
Static Two-Point Discrimination | 1.5 years
  Evaluation of sensory recovery through the measurement of the threshold of discrimination
Grip strength | 1.5 years
  Evaluation of functional recovery through the measurement of maximum grip strength
Pinch strength | 1.5 years
  Evaluation of functional recovery through the measurement of pinch strength
Patient Rated Ulnar Nerve Evaluation (PRUNE) | 1.5 years
  Evaluation of pain and quality of life through patient-reported questionnaire where lower scores indicate lower pain and better quality of life related to the injury

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No